CLINICAL TRIAL: NCT06552481
Title: A Case-Control Study of Negative Pressure Platform Wound Devices (NP-PWD) for Skin and Soft Tissue Defects
Acronym: NP-PWD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP-PWD 02
Record Dates: First submitted 2024-07-01; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Skin Wound; Soft Tissue Injuries
Keywords: Negative pressure therapy
MeSH Terms: conditions — Soft Tissue Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- NP-PWD application (Experimental): Patients randomized to NP-PWD arm will have the NP-PWD device applied to their wound.
  Interventions: Device: NP-PWD
- Standard of Care Wound VAC application (Active Comparator): Patients randomized to the standard of care arm will have the standard wound vac device applied to their wound.
  Interventions: Device: Wound Vac

INTERVENTIONS:
Device: NP-PWD — Application of NP-PWD device.
  Arms: NP-PWD application
Device: Wound Vac — Application of wound vac device.
  Arms: Standard of Care Wound VAC application

SUMMARY:
This study will demonstrate the effectiveness of the NP-PWD therapy in managing complex wounds and improving wound healing parameters as compared to standard of care.

DETAILED DESCRIPTION:
A study of 24 completed subjects will be conducted by enrolling patients who are requiring treatment for open skin and soft tissue defects. Patients will be screened for inclusion criteria and asked to consent to participate in the study. Following consent subjects will be randomized to receive treatment of one of the two study arms. Arm 1, the standard of care arm, will receive KCI Wound VAC Granulofoam. Arm 2, the study arm, will receive treatment with NP-PWD. Prior to the initial application, wound evaluations and photography will be completed to include assessment of infection with wound swabs. The wound dressing will be assessed for the need for change every 2-3 days and changed if clinically indicated (following each device IFU). Subjects will be followed for up to nine days post initial application. At minimum, the randomized treatment will be applied for 2 days after initial application for a subject to be considered completed. Subject who do not complete the treatment course (minimum of 2 days of treatment), may be replaced per investigators discretion. Follow up data will be gathered at each change/removal of the NP-PWD or Wound VAC. The data collected will include indications for dressing change, dressing change process, photographs and assessments for wound healing, infection, and adverse events. Gathered clinical data of the enrolled subjects will be used to evaluate the feasibility in using the NP-PWD device for wound healing management.

ELIGIBILITY:
Inclusion Criteria

All subjects enrolled must meet ALL the following criteria:

1. Patients 18 years of age or older of either gender
2. Have an open skin or soft tissue defect requiring treatment

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

1. Active malignant disease at the study site
2. Any concomitant medications or co-morbidities that, in the opinion of the investigator, may interfere with device use
3. On any investigational drug(s) or therapeutic device(s) to the study site in the last 30 days or any previous enrollment in this study
4. Pregnant at enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Feasibility and usability of device in treatment. | Seven to nine days post application.
  The number and type of issues with the device will be documented to determine feasibility and usability. Events such as complications with application, device changes and early removal and rationale for events during the period the patient has the study device applied and throughout the entire enrollment period.

SECONDARY OUTCOMES:
Wound readiness for closure | Seven to nine days post application.
  The treating physician will use their best medical judgment to assess the wound bed using rate of epithelization, signs of infection, exposed tendon or bone and overall appearance of the wound bed to determine the wounds readiness for closure. It will be documented the number of subjects from both groups that after treatment are ready to be grafted, or are no longer requiring surgery.
Incidence of colony forming units. | Seven to nine days post application.
  Colony forming units are assessed by obtaining wound swabs and analysis of presence of colony forming units.
Ease of use of device by healthcare providers | Seven to nine days post application.
  At each research visit the staff will be asked if they had any questions, concerns, complaints or comments about the device or dressing. There is not a separate healthcare provider questionnaire, but any information obtained will be placed in the comments section of the source documents and the feedback will be provided to manufacture.
Tolerability of the device by patient subjects | Seven to nine days post application.
  Tolerability of device by subjects will be assessed by observation of the length of time subjects were able to keep the dressing on. The subject will be asked if they have any concern or complaints about the device or dressing. Their response and if applicable the reason for removal will all be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Chan, MD, Principal Investigator — The Metis Foundation
Locations (1):
- Northeast Baptist, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT06552481/Prot_SAP_000.pdf